CLINICAL TRIAL: NCT01226238
Title: Online Self-help for Depressed Patients Awaiting Psychotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Philipp Klein, Dr. med., University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Deprexis-HH-HL-WL
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Online self-help (Experimental): Provision of online self-help while waiting for psychotherapy
  Interventions: Other: Online self-help
- Waiting list alone (No Intervention): Waiting for psychotherapy alone

INTERVENTIONS:
Other: Online self-help — Provision of online self-help
  Arms: Online self-help

SUMMARY:
Patients with major depression who are on a waiting list for psychotherapy usually suffer from considerable symptoms. Online self-help is one potential way to alleviate this suffering. The investigators want to study if patients awaiting psychotherapy benefit from online-self help. The investigators therefore randomly assign patients to either online self-help or no intervention and assess their depressive symptoms on a regular basis. The investigators hypothesize that online self-help will be superior to no intervention in alleviating depressive symptoms in depressed patients awaiting psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder
* stable medication
* 18yrs. or older

Exclusion Criteria:

* current psychotherapy
* acute suicidality
* unavailability of internet connection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Depressive Symptomatology | up to 16 weeks

SECONDARY OUTCOMES:
Depressive Symptomatology | 6 weeks, up to 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- MVZ Falkenried, Hamburg, Germany

REFERENCES:
- [Derived] Klein JP, Roniger A, Schweiger U, Spath C, Brodbeck J. The association of childhood trauma and personality disorders with chronic depression: A cross-sectional study in depressed outpatients. J Clin Psychiatry. 2015 Jun;76(6):e794-801. doi: 10.4088/JCP.14m09158. PMID 26132688